CLINICAL TRIAL: NCT00223509
Title: Lamictal As Add on Treatment in Mixed States of Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0340013418
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Bipolar Disorder
Keywords: mixed mania; lamotrigine
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lamotrigine

SUMMARY:
* To evaluate the efficacy and safety of LAM+existing regimen of mood stabilizer in the acute treatment of patients in a mixed state of bipolar disorder.
* To evaluate the efficacy and of a combination of LAM+existing regimen of mood stabilizers in the maintenance treatment of patients with mixed state of bipolar disorder

DETAILED DESCRIPTION:
1. To evaluate the efficacy and safety of LAM+existing regimen of mood stabilizer in the acute treatment of patients in a mixed state of bipolar disorder.
2. To evaluate the efficacy and of a combination of LAM+existing regimen of mood stabilizers in the maintenance treatment of patients with mixed state of bipolar disorder

ELIGIBILITY:
Inclusion Criteria:

In order to be included in the study patient must meet criteria A, C, D, E, F, G plus any 1 of the 3 criteria listed in section B.

A. Patients meeting DSM-IV diagnosis of bipolar disorder, I or II

B.

1. Patients meeting DSM-IV diagnostic criteria for a manic/hypomanic episode with the simultaneous presence of (or rapid alteration within minutes) of at least three DSM-IV depressive symptoms excluding psychomotor agitation or
2. Patients meeting DSM-IV symptomatic criteria for a hypomanic/manic episode for a period of 2 days or longer, with the simultaneous presence of (or rapid alteration within minutes) of at least three DSM-IV depressive symptoms excluding psychomotor agitation or
3. Patients meeting DSM-IV criteria for a depressive episode associated with at least three DSM-IV manic/hypomanic symptoms

C.MADRS of ≥14

D.YMRS of ≥ 14

E. Age 13years to 75 years

F. Male or female

G. Outpatient

Exclusion Criteria:

1. illness precluding the use of LAM
2. Alcohol/drug dependence in the past one month
3. patients with a history of a rash on LAM
4. CNS neoplasms, demyelinating diseases, degenerative neurological condition or active CNS infection
5. history of seizure, known EEG with frank paroxysmal activity, known CT of brain showing gross structural abnormalities, cerebral vascular disease by history or structural brain damage from trauma
6. patients currently taking LAM

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Primary efficacy, during the first 10 weeks (acute phase) of the study, will be assessed by the proportion of patients achieving a 50% reduction of their depressive symptoms as assessed by the MADRS and a GAF | 12 weeks
MADRS | 12 weeks
Efficacy, during the maintenance phase of the study, will be assessed by the proportion of patients able to maintain a response, at the end of the study, as defined by
MADRS total score of <14, GAF score 51. Secondary measures will include the YMRS, and CGI Bipolar version.

SECONDARY OUTCOMES:
Secondary measures will include the YMRS, and CGI Bipolar version.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek - Singh, MD, Principal Investigator — University of Texas; Charles L Bowden, MD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - Univ of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas